CLINICAL TRIAL: NCT00777712
Title: Mechanisms Underlying Impaired Diabetic Wound Healing
Acronym: WoundVac
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sashwati Roy, Professor, University of Pittsburgh
Other Study IDs: STUDY23070132
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Non-healing Wounds; Diabetes
Keywords: Wound healing; diabetes; inflammatory cell; monocyte; leukocyte; macrophage
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Wound Vac Sponge.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic wound study: Patients with diabetes or no diabetes
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood will be drawn from subjects once and VAC sponge will be collected (which is normally discarded material per standard of care).

SUMMARY:
The overall aim of this research is to utilize wound derived inflammatory cells from diabetic versus non diabetic human chronic wounds to understand mechanisms that are responsible for disregulated inflammation in individuals with diabetes. Biology of normal (peripheral blood derived cells) versus wound derived cells will also be studied.

DETAILED DESCRIPTION:
Specific aims:

1. To study biology of wound derived inflammatory cells and fluid from diabetic versus non diabetic wounds.
2. To characterize mechanisms that are responsible for dysregulated wound inflammatory cell function in individuals with diabetes.
3. To characterize differences in the biology of normal peripheral blood derived cells versus wound derived cells.

The long-term goal of this study is to determine the molecular mechanisms underlying impaired wound healing in diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-80
* Chronic Wound (present >4 weeks)
* Diabetic & Non-diabetic
* Adult surgical wounds

Exclusion Criteria:

* Inability to consent
* Pregnant women
* Therapeutically immunocompromised
* Individuals defined in 45 CFR 46 Subparts B,C, and D, nor from any other population considered vulnerable 2.9

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Comprehensive Wound Care Centers: Indiana University/ Indiana University Health Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing | Week 16
  Wound healing status

SECONDARY OUTCOMES:
Infection status | week 0
  CFU analysis of the wound fluid

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, Ph.D., Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Comprehensive Wound Care Centers, Indianapolis, Indiana
  - Comprehensive Wound Care Centers, Columbus, Ohio
  - University of Pittsburgh - McKeesport, Pittsburgh, Pennsylvania
  - University of Pittsburgh - Mercy, Pittsburgh, Pennsylvania
  - University of Pittsburgh - Passavant, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Mousley M. Diabetes and its effect on wound healing and patient care. Nurs Times. 2003 Oct 21-27;99(42):70, 73-4. PMID 14618996
- [Background] Stadelmann WK, Digenis AG, Tobin GR. Impediments to wound healing. Am J Surg. 1998 Aug;176(2A Suppl):39S-47S. doi: 10.1016/s0002-9610(98)00184-6. PMID 9777971
- [Background] Meehan M, O'Hara L, Morrison YM. Report on the prevalence of skin ulcers in a home health agency population. Adv Wound Care. 1999 Nov-Dec;12(9):459-67. PMID 10687558
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2007 Jan;30 Suppl 1:S42-7. doi: 10.2337/dc07-S042. No abstract available. PMID 17192378
- [Background] American Diabetes Association. Standards of medical care in diabetes--2007. Diabetes Care. 2007 Jan;30 Suppl 1:S4-S41. doi: 10.2337/dc07-S004. No abstract available. PMID 17192377
- See also: IU Center for Regenerative Medicine and Cell Based Therapies — https://medicine.iu.edu/research-centers/regenerative-medicine-engineering